CLINICAL TRIAL: NCT00605085
Title: Safety and Tolerability of the Japanese Encephalitis Vaccine IC51. Double Blind, Randomized, Placebo Controlled Phase 3 Study
Brief Title: Safety and Tolerability of the Japanese Encephalitis Vaccine IC51
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Intercell AG
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IC51-302
Record Dates: First submitted 2008-01-04; First posted 2008-01-30 (Estimated); Results first posted 2012-11-20 (Estimated); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): IC51
  Interventions: Biological: Japanese Encephalitis purified inactivated vaccine (IC51)
- 2 (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Japanese Encephalitis purified inactivated vaccine (IC51) — IC51 (JE-PIV), 6 mcg, i.m. injection, 2 vaccinations, days 0 and 28
  Arms: 1
Biological: Placebo — Placebo: Phosphate-buffered saline (PBS) solution containing 0.1% aluminum hydroxide as an adjuvant, 0.5 mL, i.m. injection, 2 injections, days 0 and 28
  Arms: 2

SUMMARY:
The objective is to investigate the safety and tolerability of Japanese Encephalitis vaccine IC51 with an inactive control in healthy subjects aged > or = 18 years

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Written informed consent obtained prior to study entry

Exclusion Criteria:

* Use of any other investigational or non-registered drug or vaccine in addition to the study vaccine during the study period or within 30 days preceding the first dose of study vaccine
* History of any previous JE vaccination (e.g. JE-VAX®)
* Immunodeficiency including post-organ-transplantation or immunosuppressive therapy
* A family history of congenital or hereditary immunodeficiency
* History of autoimmune disease
* Any acute infections within 2 weeks prior to enrollment
* Known or suspected HIV Infection
* Pregnancy, lactation or unreliable contraception in female subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2675 (Actual)
Dates: Start 2005-10; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Kaltenboeck, Ph.D., Study Director — Valneva Austria GmbH

RESULTS

PARTICIPANT FLOW:
Groups:
- IC51: IC51
- Placebo: Placebo
Period: Overall Study
Arm/Group | IC51 | Placebo
Started | 2012 | 663
Completed | 1962 | 638
Not Completed | 50 | 25
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Adverse Event | 9 | 5
Not completed — Pregnancy | 2 | 0
Not completed — Protocol Violation | 3 | 2
Not completed — Lost to Follow-up | 10 | 5
Not completed — administrative reasons | 18 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IC51 | Placebo | Total
Number analyzed (Participants) | 1993 | 657 | 2650
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (13.3) | 33.4 (13) | 33.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1088 | 378 | 1466
  Male | 905 | 279 | 1184
Region of Enrollment [Number; unit: participants]
  Australia | 294 | 100 | 394
  Europe | 1236 | 406 | 1642
  United States | 463 | 151 | 614

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability up to Day 56
Description: calculation based on safety population, numbers provide percentages of participants with Adverse Events (AEs)
Time Frame: Day 56
Population: Safety Population
Measure: Number; unit: percentage of participants with AEs
Arm/Group | IC51 | Placebo
Number analyzed (Participants) | 1993 | 657
percentage of participants with AEs | 58.9 | 56.6

2. Secondary Outcome: Rates of Serious Adverse Events and Medically Attended Adverse Events
Time Frame: until Day 56
Reporting Status: Not Posted

3. Secondary Outcome: Changes in Laboratory Parameters
Time Frame: until Day 56
Reporting Status: Not Posted

4. Secondary Outcome: SCR and GMT of Subjects With Concomitant Vaccinations
Time Frame: until Day 56
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Safet population (N = 2650): All subjects who entered the study and received at least one vaccination. All analyses based on the safety population were carried out using the actual treatment received.
  The safety population was used for all safety and tolerability analyses and for the analysis of demographic and background data.
Arm/Group | IC51 | Placebo
Serious Adverse Events (participants affected / at risk) | 10/1993 | 6/657
Other Adverse Events (participants affected / at risk) | 917/1993 | 292/657
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IC51 (N=1993) | Placebo (N=657)
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Abscess Limb (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 2
Face Injury (Injury, poisoning and procedural complications) | 1 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0
Ulna Fracture (Injury, poisoning and procedural complications) | 1 | 0
Calculus Urinary (Renal and urinary disorders) | 0 | 1
Adnexa Uteri Pain (Reproductive system and breast disorders) | 1 | 0
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 1 | 0
Ovarian Torsion (Reproductive system and breast disorders) | 1 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 | 0
Curculatory Collapse (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IC51 (N=1993) | Placebo (N=657)
Nausea (Gastrointestinal disorders) | 131 | 49
Fatigue (General disorders) | 227 | 77
Influenza Like Illness (General disorders) | 248 | 78
Pyrexia (General disorders) | 64 | 20
Nasopharyngitis (Infections and infestations) | 94 | 26
Myalgia (Musculoskeletal and connective tissue disorders) | 311 | 102
Headache (Nervous system disorders) | 559 | 173

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other